CLINICAL TRIAL: NCT07324850
Title: A Phase 1, Randomized, Double-blind, Placebo-controlled Single Ascending Dose Study to Evaluate the Safety, Tolerability, Pharmacokinetics, and Pharmacodynamics of Subcutaneously Administered SGB-7342 in Subjects With Obesity or Overweight
Brief Title: A Study of SGB-7342 in Subjects With Obesity or Overweight
Status: Not yet recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Suzhou Sanegene Bio Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SGB-7342-001
Record Dates: First submitted 2025-12-23; First posted 2026-01-08 (Actual); Last update posted 2026-01-09 (Actual); Status verified 2026-01

CONDITIONS: Obesity & Overweight
MeSH Terms: conditions — Obesity; Overweight

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- SGB-7342 (Experimental)
  Interventions: Drug: SGB-7342
- SGB-7342-Matching placebo (Placebo Comparator)
  Interventions: Drug: SGB-7342-Matching placebo

INTERVENTIONS:
Drug: SGB-7342 — SC injection, single dose
  Arms: SGB-7342
Drug: SGB-7342-Matching placebo — Normal saline (0.9% NaCl) in a matching volume, SC injection, single dose
  Arms: SGB-7342-Matching placebo

SUMMARY:
The purpose of this study is to evaluate the safety and tolerability of subcutaneously administered SGB-7342 in adult subjects with obesity and overweight.

ELIGIBILITY:
Inclusion Criteria:

* Body Mass Index (BMI) within the range of 26.0 to 35.0 kg/m²
* Have a stable body weight within 3 months
* Participants must agree to use adequate contraception from signing the informed consent until 6 months after completion of the follow-up visit.
* Willing to comply with the protocol required visit schedule and visit requirements and provide written informed consent.

Exclusion Criteria:

* A history of or a current surgical or medical condition that, in the opinion of the Investigator, may put the subject at significant risk (according to Investigator's judgment) or interfere with the subject's participation in the clinical study.
* Use of GLP-1R agonists for any indication within 6 months prior to administering the investigational drug.
* Use of non-GLP1R medications for weight loss within 3 months prior to administering the investigational drug.
* Alanine aminotransferase (ALT), total bilirubin (TBIL), aspartate aminotransferase (AST)> 1.5 × ULN, and deemed clinically significant by the Investigators

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 45 (Estimated)
Dates: Start 2026-01-12 (Estimated); Primary Completion 2026-10-28 (Estimated); Study Completion 2027-04-14 (Estimated)

PRIMARY OUTCOMES:
Number of Participants with Adverse Events (AEs) | up to approximately 6 months

SECONDARY OUTCOMES:
Maximum Observed Plasma Concentration (Cmax) | up to approximately 3 days
Area Under the Concentration-time Curve (AUC) | up to 3 days
Weight change from baseline | up to approximately 12 months